CLINICAL TRIAL: NCT04694040
Title: Analysis of Mandibular Kinematics of a Group of Asymptomatic Subjects Recorded With the Modjaw® Device
Brief Title: Condylar Inclination Recorded With Modjaw® Device.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20odonto01
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy adult volunteers showing no signs of temporomandibular disorders
  Interventions: Device: Modjaw® device

INTERVENTIONS:
Device: Modjaw® device — Analysis of mandibular kinematics with Modjaw® device

SUMMARY:
In oral rehabilitation, the integration into the digital flow of mandibular movements and the patient's individual reference planes optimizes the functional adaptation of prosthetic elements whose design is computer aided. The innovative Modjaw® device allows you to record and then virtually simulate mandibular movements.

This retrospective study aims to: 1) Test the reliability of the Modjaw® device; 2) Measure the condylar displacements of asymptomatic subjects for the arbitrary programming of simulators.

Kinematic recordings of 22 healthy volunteers (15F / 7H; mean age: 22.2 years) were analyzed. Two recording sessions were carried out within one month of each other, by three different operators; each subject was followed by the same operator during the first (E1) and the second (E2) recording. The values of sagittal condylar inclination (SCI) obtained in opening, protrusion, right-left mediotrusion were calculated at 3 and 5 mm of condylar displacement. The transverse condylar inclination (TCI) was calculated at 4mm.

ELIGIBILITY:
Inclusion criteria : adult ;

Exclusion criteria : temporomandibular disorders (TMD symptom questionnaire)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Reliability of recordings | 5 months
  The intra-class correlation coefficient (ICC) based on a one-way random-effects ANOVA was used to measure the repeatability of the recordings.

SECONDARY OUTCOMES:
Mandibular motion | 5 months
  Sagittal and transversal condylar inclination mesured in degrees

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE - Hôpital St Roch, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing is planned